CLINICAL TRIAL: NCT05605587
Title: Leflunomide Treatment for MEN1 Patients - the LUMEN1 Trial
Acronym: LUMEN1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was prematurely terminated due to significant difficulties in recruiting participants, arising from the extremely rare nature of the targeted gene mutation.
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUMEN1
Record Dates: First submitted 2022-11-01; First posted 2022-11-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: MEN1 Gene Mutation
MeSH Terms: interventions — Leflunomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Leflunomide 20mg (Experimental)
  Interventions: Drug: Leflunomide 20 mg

INTERVENTIONS:
Drug: Leflunomide 20 mg — once daily for 6 months

SUMMARY:
Multiple endocrine neoplasia type 1 (MEN1) is an autosomal dominant disorder due to mutations in the tumor suppressor gene MEN1 with the corresponding gen product menin. MEN1 is characterized by the occurrence of parathyroid, pancreatic islet and anterior pituitary tumors which can release excessive amounts of hormones (= functional active tumors). Other tumors (e.g. carcinoid tumors, adrenocortical tumors, meningiomas, facial angiofibromas, collagenomas, lipomas) have also been described. There is no geno-phenotype correlation but the disease occurs after a second hit of the corresponding gene within the endocrine organ leading to an uncontrolled growth.

MEN1-patients have a decreased life expectancy, mainly due to pancreatic neuroendocrine tumors (pNETs) which are often multiple and more aggressive than in non-MEN1 patients. To date, no prophylactic treatment exists to prevent tumor development in this hereditary disease.

Leflunomide has been used as a treatment for rheumatoid arthritis for many years. It is a potent inhibitor of the dihydroorotate dehydrogenase (DHODH). According to some preclinical studies, leflunomide showed antineoplastic activities in several malignancies, including prostate, breast, bladder, multiple myeloma, leukemia, and lymphoma. A recent study identified an interaction between MEN1 mutation and DHODH inhibition. In this study, leflunomide selectively killed MEN1 deficient cells in vitro, prevented the occurrence of pancreatic tumor development in xenograft models and led to tumor regression / stabilisation in three MEN1 patients with advanced aggressive pancreatic neuroendocrine tumors.

Accordingly, leflunomide could be used as a new treatment option for patients with known MEN1 germline mutation and associated endocrine disease. The aim of this study is, therefore, to evaluate the antitumor effect of leflunomide treatment on MEN1-associated tumors in patients with known MEN1-syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) patients with known pathogenic or likely pathogenic MEN1-germline mutation and at least 1 associated tumor lesion OR hormonal syndrome

Exclusion Criteria:

* uncontrolled arterial hypertension, defined as blood pressure >160/100 mmHg
* Impaired kidney function, defined as creatinine clearance <50ml/min
* Impaired liver function, defined as bilirubin or liver transaminases >3 times upper normal range
* Cytopenia, defined as one or several of the following: hemogloin <100 g/l, leucopenia <2x109/l, thrombocytopenia <100x109/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2026-01-13 (Actual); Study Completion 2026-01-13 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the effect of a 6 months' treatment with leflunomide 20mg/day on MEN1-associated functional and non-functional tumors | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Unispital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided